CLINICAL TRIAL: NCT07163403
Title: First in Human Pilot Study to Assess the Safety and Efficacy of Dendritic Cells Loaded With Frameshift Derived Neopeptides for the Prevention of Cancer in of Lynch Syndrome Carriers
Acronym: DELAY
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2025-521109-42-00
Record Dates: First submitted 2025-07-30; First posted 2025-09-09 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Lynch Syndrome
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Patients with Lynch Syndrome which will recieve their own dendritic cells to evaluate safety and tolerability
  Interventions: Biological: Autologous Tolerogenic Dendritic cells

INTERVENTIONS:
Biological: Autologous Tolerogenic Dendritic cells — Autologous peripheral blood differentiated and matured adult dendritic cells loaded with Frameshift-derived neopeptides (FSDN) (DC-DELAY). Eligible participants will receive six intradermal immunizations of DC-DELAY at week 0, 2, 4, 6, 8 and 10.

SUMMARY:
Tha aim of this clinical trial is to evaluate safety and tolerability of autologous peripheral blood differentiated and matured adult dendritic cells. Immunogenicity of the prduct(DC-DELAY) will be evaluated also.

DETAILED DESCRIPTION:
First in human, pilot, open-label, prospective, single-site, non-randomised study

ELIGIBILITY:
Inclusion Criteria:

1. Individuals that are carriers of a pathogenic or likely pathogenic germline variant in one of the mismatch repair genes (MLH1, MSH2, MSH6).
2. Participants must have no evidence of active or previous invasive cancer.
3. Participants must have endoscopically accessible colon.
4. Participants must consent to follow the standard of care surveillance with colonoscopy and biopsies every 1-2 years.
5. Age ≥ 18 years
6. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1 (Karnofsky ≥70%).
7. Haemoglobin ≥10 g/dL or haematocrit ≥30%; Leukocyte count ≥3.0x109/l; Platelet count ≥100x109/l; Absolute neutrophil count ≥1.5x109/l; Absolut lymphocyte count ≥0.8x109/l.
8. Creatinine clearance (calculated if measured is not available) ≥60mL/min/1.73m2.
9. Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT] ≤2 times the institutional upper limit of normal (ULN).
10. Total bilirubin ≤ 1.5 the ULN; participants with Gilbert's disease may be enrolled with higher total bilirubin if their direct bilirubin is ≤1.5 times the ULN.
11. Written informed consent.
12. Women of child-bearing potential* must have a negative pregnancy test in serum before the inclusion in the study and agree to use highly effective contraceptive methods until one year following the las immunization dose. Highly effective contraceptive methods will include: combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable), intrauterine device, bilateral tubal occlusion, vasectomized partner and sexual abstinence. * A woman will be considered of childbearing potential, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A postmenopausal state is defined as 0 menses for 12 months without an alternative medical cause. A high follicle stimulating hormone level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single follicle stimulating hormone measurement is insufficient.

Exclusion Criteria:

1. Individuals that are carriers of a pathogenic or likely pathogenic germline variant in PMS2.
2. Individuals with active malignancy or previous malignancy (excluding non-melanoma skin cancer)
3. Participants who cannot be removed from their baseline medication for the duration of the trial to administer the investigational treatment. This includes the daily use of >100 mg aspirin or nonsteroidal anti-inflammatory drugs (NSAIDs) or cyclooxygenase (COX) inhibitors.
4. Any serious uncontrolled and /or unstable pre-existing medical disorder (aside from malignancy exception above), psychiatric disorder, or other conditions that could interfere with participant's safety, obtaining informed consent, or compliance to the study procedures.
5. Patients with active systemic bacterial, viral or fungal infections or known to have human immunodeficiency virus (HIV) or to test positive for HIV antibody at screening.
6. Positive hepatitis B surface antigen or hepatitis C antibody tests at screening.
7. History of organ allograft or other history of immunodeficiency
8. Individuals with a condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications.
9. Pregnant or breastfeeding or planning to become pregnant during the first year after the completion of the study treatment.
10. Men attempting or planning to conceive children during the first year after the completion of the study treatment.
11. Participants cannot receive any other investigational agents in the last month before its inclusion.
12. Participants unable to refrain to receive any type of vaccination during the first 12 weeks of the trial.
13. Impossibility to proceed to the leukapheresis (e.g. absence of peripheral venous access).
14. Any other problem that according to the investigator could interfere with the evaluation of the objectives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-04 (Actual); Primary Completion 2028-09-20 (Estimated); Study Completion 2028-09-20 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with grade 3-4 related adverse events for 12 months following the first immunization. | the first 12 month after the last inmunization
  To evaluate the safety and tolerability of autologous peripheral blood differentiated and matured adult dendritic cells loaded with frameshift derived neopeptides (DC-DELAY) in LS carriers.
Proportion of participants with specific frameshift-derived neoantigens immune response induced by DC-DELAY as measured in peripheral blood by enzyme-linked immune absorbent spot(ELISpot) assay at week 12. | At week 12.
  To evaluate specific frameshift-derived neoantigens immunogenicity of DC-DELAY in LS carriers at week 12. NOTE: Immune response will be defined as T-cell reactivity to at least 1 out of 4 of the pools.

SECONDARY OUTCOMES:
Proportion of participants with early immune response induced by DC-DELAY as measured inperipheral blood by ELISpot assay at week 6. | Week 6
  To evaluate the early-term specific frameshift-derived neoantigens immunogenicity of DC-DELAY in LS carriers at week 6.
Proportion of participants with long term immune response induced by DC-DELAY as measured in peripheral blood by ELISpot assay at months 6, 12 and 24. | Month 6, 12 and 24.
  To evaluate the long-term specific frameshift-derived neoantigens immunogenicity of DC-DELAY in LS carriers at 6, 12 and 24 months.
Proportion of participants with immune response induced by DC-DELAY as measured in the normal colonic mucosa at month 12. | Month 12
  To evaluate the specific frameshift-derived neoantigens immunogenicity of DC-DELAY in the normal colonic mucosa in LS carriers at month 12.
Proportion of participants with mismatch repair deficient colorectal adenomas, advanced neoplasia and/or carcinoma throughout the study duration. | Month 12 and month 36
  To evaluate the effect of DC-DELAY in LS carriers at week 12 on the burden of mismatch repair deficient colorectal neoplasia throughout the study duration.
Proportion of participants with LS-related carcinomas throughout the study duration (36 months). | Week 12 and month 36
  To evaluate the effect of DC-DELAY immunization in LS carriers at week 12 on the burden of LSrelated carcinomas throughout the study duration.
Number and proportion of participants with related adverse events at 7 days after each DC-DELAY immunization. | 7 days after each iminization, week 0, week 2, week 4, week 6, uweek 8 and week 10.
  To evaluate the safety and tolerability of DC-DELAY
Number and proportion of participants with grade 3-4 related adverse events throughout the study duration (36 months). | Through study completion, an average of 3 years.
  To evaluate the safety and tolerability of DC-DELAY throughout the study duration.

CONTACTS AND LOCATIONS:
Locations (1):
- Laura Burunat, Barcelona, Barcelona, Spain